CLINICAL TRIAL: NCT07075770
Title: Novel Personalized Non Invasive Combined Magnetic and Electrical Stimulation of the Default Mode Network in Mild AD Patients (CMES-AD)
Brief Title: Novel Personalized Non Invasive Combined Magnetic and Electrical Stimulation of the DMN in Mild AD Patients
Acronym: CMES_AD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PNRR-MCNT2-2023-12377518
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease
Keywords: Non Invasive Brain Stimulation; Transcranial Magnetic Stimulation; Intermittent Theta Burst Stimulation; Transcranial Electrical Stimulation; Transcranial Alternating Current Stimulation; Default Mode Network
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Three arms randomized sham-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Four-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- combined iTBS-tACS (Experimental): 32 sessions of combined iTBS-tACS (5 times/week for 2 weeks -intensive phase-; 1 time/week for 22 weeks -maintenance phase-)
  Interventions: Device: Combined iTBS-tACS
- iTBS-sham tACS (Active Comparator): 32 sessions of combined iTBS-sham tACS (5 times/week for 2 weeks -intensive phase-; 1 time/week for 22 weeks -maintenance phase-)
  Interventions: Device: iTBS-sham tACS
- sham iTBS- sham tACS (Placebo Comparator): 32 sessions of sham iTBS- sham tACS (5 times/week for 2 weeks -intensive phase-; 1 time/week for 22 weeks -maintenance phase-)
  Interventions: Device: sham iTBS- sham tACS

INTERVENTIONS:
Device: Combined iTBS-tACS — The iTBS-tACS will be applied over the precuneus and last for 190 s, with the tACS electrode positioned on the scalp and the iTBS coil positioned just above it. The iTBS protocol will consist of 600 pulses, delivered in 20 trains of 10 bursts with an interval of 8 seconds between each train. Each burst consists of three pulses at 50Hz, repeated at 5Hz. The total duration will therefore be 190 seconds. iTBS and tACS will be synchronized using a BrainTrigger and SIGNAL Software so that both stimulations will start simultaneously
  Arms: combined iTBS-tACS
Device: iTBS-sham tACS — The iTBS-tACS will be applied over the precuneus and last for 190 s, with the tACS electrode positioned on the scalp and the iTBS coil positioned just above it. The iTBS protocol will consist of 600 pulses, delivered in 20 trains of 10 bursts with an interval of 8 seconds between each train. Each burst consists of three pulses at 50Hz, repeated at 5Hz. The total duration will therefore be 190 seconds.
  For the tACS sham condition, the electric current will not be applied, but there will be a 2 s 1 mA ramp up and 2 s 1 mA ramp down, to give the participant real stimulation feelings.
  Arms: iTBS-sham tACS
Device: sham iTBS- sham tACS — The iTBS-tACS will be applied over the precuneus and last for 190 s, with the tACS electrode positioned on the scalp and the iTBS coil positioned just above it. The iTBS protocol will consist of 600 pulses, delivered in 20 trains of 10 bursts with an interval of 8 seconds between each train. Each burst consists of three pulses at 50Hz, repeated at 5Hz. The total duration will therefore be 190 seconds.
  For the iTBS sham condition, stimulation was delivered with the coil angled at 90°, with only the edge of the coil resting on the scalp..
  For the tACS sham condition, the electric current will not be applied, but there will be a 2 s 1 mA ramp up and 2 s 1 mA ramp down, to give the participant real stimulation feelings.
  Arms: sham iTBS- sham tACS

SUMMARY:
Alzheimer's disease (AD) is increasingly recognized as a disorder marked by early synaptic dysfunction and disrupted brain network connectivity, beyond the traditional focus on amyloid pathology. Synaptic plasticity (crucial for learning and memory) is compromised in AD and represents a promising therapeutic target. In particular, alterations in the Default Mode Network (DMN), especially in regions like the precuneus, suggest that restoring connectivity and enhancing plasticity may improve cognitive outcomes. This project proposes a novel, precision-delivered non-invasive brain stimulation protocol that combines repetitive transcranial magnetic stimulation (rTMS) and transcranial alternating current stimulation (tACS) over the DMN. The intervention will be evaluated through cognitive testing, blood-based biomarkers, MRI and TMS-EEG, alongside immersive virtual environments to assess sensorimotor and cognitive function. This approach aims to test neuromodulation strategies capable of slowing neurodegeneration and supporting early detection and rehabilitation in AD.

DETAILED DESCRIPTION:
Patients will be screened at trial sites for determination of eligibility to enter the study on the basis of diagnostic evaluations, according to current diagnostic criteria for probable AD, and safety assessments (vital sign complete physical and neurological examinations). The efficacy assessments (cognitive/behavioral evaluations) will be performed at Baseline before starting treatment and repeated on- treatment at Weeks 0, 12 and 24. Plasma biomarkers will be collected at baseline and at Week 12 and 24. Visit windows are ±7 days for all the scheduled visits. In case a visit is performed outside its window, subsequent visits will be performed in keeping with the original visit schedule. At each in-clinic visit (or upon early termination), AEs will be recorded, at screening, baseline, Week 12 and 24 vital signs measured, and physical and neurological examination performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of AD according to IWG criteria
* 20 > MMSE < 28
* Patients with CSF specific biomarker profile or with a positive Amyloid Pet Scan consistent with the presence of amyloid pathology
* Global Clinical Dementia Rating (CDR) ≤1
* Previous decline in cognition for more than six months as documented in patient medical records
* A caregiver available and living in the same household or interacting with the patient and available
* Patients living at home or nursing home setting without continuous nursing care
* General health status acceptable for a participation in a 6-month clinical trial
* Stable pharmacological treatment for at least one month prior to screening
* No regular intake of prohibited medications.
* Signed informed consent by the patient. If there are any doubts that the patient is mentally capable of giving informed consent, the patient will be examined and verified to be mentally capable by an independent physician/ neurologist, prior to the initiation of any study specific procedure. Signed consent of the caregiver

Exclusion Criteria:

* Failure to undergo screening or baseline exams
* Hospitalization or change in chronic concomitant medications one month before the screening or during the screening period
* Clinical, laboratory, or neuroimaging results consistent with:

  1. other primary degenerative dementia (Lewy body dementia, frontotemporal dementia, Huntington's disease, Creutzfeldt-Jakob disease, Down syndrome, etc.);
  2. other neurodegenerative conditions (Parkinson's disease, amyotrophic lateral sclerosis, etc.);
  3. orthostatic hypotension and autonomic disorders
  4. cerebrovascular disease (major infarction, a strategic infarction or multiple lacunar infarctions, extensive white matter lesions > one quarter of total white matter);
  5. other central nervous system diseases (severe traumatic brain injury, tumors, subdural hematoma, or other space-occupying processes, etc.);
  6. seizure disorder.
  7. Other infectious, metabolic, or systemic diseases affecting the central nervous system (syphilis, existing hypothyroidism, current vitamin B12 or folate deficiency, serum electrolytes outside normal limits, juvenile diabetes, etc.).
* A current DSM-V diagnosis of major depression, schizophrenia, or bipolar disorder.
* Clinically significant, advanced, or unstable disease that may interfere with primary or secondary variable assessments and may affect the assessment of the patient's clinical or mental state, or expose the patient to special risk, such as:

  1. Disability that may prevent the patient from completing all study requirements (e.g., blindness, deafness, severe language difficulties, etc.);
  2. Opioid-containing analgesics
  3. Suspected or known drug or alcohol abuse, i.e., more than about 60 g of alcohol (about 1 liter of beer or 500 ml of wine) per day, indicated by a high mean corpuscular volume (MCV) above the normal value at screening;
  4. Any condition that, in the investigator's judgment, makes the patient unsuitable for inclusion

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
integrated Alzheimer Disease Rating Scale (iADRS) | Change from baseline to the end of treatment at week 24.
  The iADRS is an integrated assessment of cognition and daily function from the 13-item cognitive subscale of the Alzheimer Disease Assessment Scale (ADAS-Cog13) and Alzheimer Disease Cooperative Study-Instrumental Activities of Daily Living (ADCS-iADL), measuring global disease severity across the Alzheimer disease continuum as a single summary score. The iADRS is validated and captures clinical progression from MCI due to Alzheimer disease through moderate dementia due to Alzheimer disease, and treatment effects have been demonstrated across MCI and Alzheimer disease with mild dementia. The possible scores on the iADRS range from 0 to 144 (lower scores indicate greater impairment).

SECONDARY OUTCOMES:
Change in the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) score. | Change from baseline to the end of treatment at week 24.
  The ADCS-ADL includes 23 items that were derived from a larger set of items describing performance of activities of daily living.
Alzheimer Disease Cooperative Study-Instrumental Activities of Daily Living (ADCS-iADL). | Change from baseline to week 24.
  A standardized clinical scale used to assess an individual's ability to perform complex daily tasks.
Change in the Clinical Dementia Rating scale Sum of Boxes (CDR-SoB) score. | Change from baseline to the end of treatment at week 24.
  The CDR-SoB is a 5-point scale used to characterize six domains of cognitive and functional performance in AD and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care.
Change in the Alzheimer Disease Assessment Cognitive Scale (ADAS-Cog13) score. | Change from baseline to the end of treatment at week 24.
  The ADAS-Cog13 assesses the level of cognitive function in Alzheimer's Disease. The ADAS-Cog13 consists of items from the following areas chosen for their sensitivity to Alzheimer's Disease: language; memory; praxis executive functions and orientation.
Change in the Neuropsychiatric Personal Inventory (NPI) score. | Change from baseline to the end of treatment at week 24.
  The NPI scale assesses behavioral disturbances in dementia. The NPI is a reliable and valid scale measuring the following behavioral areas: delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability, aberrant motor behavior, night time behaviors, and eating disorders. The score range is from 0 to 144 with the higher score meaning more severe behavioural disturbances.
Change in the Mini-Mental State Examination (MMSE) score. | Change from baseline to the end of treatment at week 24.
  The MMSE is a brief, widely used valid, and reliable assessment of cognitive impairment. This 30-point questionnaire is used to screen and estimate the severity of cognitive impairment in addition to being used to follow the course of cognitive change over time. The test assesses orientation, attention and calculation, recall, language, repetition, and ability to follow complex commands. The score range is from 0 to 30, with lower score meaning greater cognitive impairment.
Change in the Montreal Overall Cognitive Assessment (MoCA) score. | Change from baseline to the end of treatment at week 24.
  The MoCA is a brief screening tool for mild cognitive impairment, scored from 0 to 30, with higher scores indicating better cognitive functions.
Change in Face-Name Association Task (FNAT) score. | Change from baseline to the end of treatment at week 24.
  The FNAT is a cross-modal memory test where participants learn and recall pairs of unfamiliar faces and common first names. In this study, only face-name pairs were used (no occupations). The score reflects the number of correctly recalled names, with higher scores indicating better associative memory.
Change in Apathy Motivation index (AMI) score. | Change from baseline to the end of treatment at week 24.
  The AMI scores range from 0 to 4 for each item, with higher scores indicating greater levels of apathy. The total score is calculated by averaging item scores across its subscales.
Change in the Frontal Assessment Battery (FAB) score. | Change from baseline to the end of treatment at week 24.
  The FAB is a brief battery of six neuropsychological tasks designed to assess frontal lobe function.

OTHER OUTCOMES:
Change in cortical activity | Change from baseline to the end of treatment at week 24.
  From TMS-EEG recording it is possible to analyze oscillatory activity of the stimulated brain area. Monitoring the frequency band during time after TMS-pulse we calculate Time-frequency Wavelets and from there the TMS-related spectral perturbation (TRSP) as output of the frequency bands (Delta, Theta, Alpha, Beta, Gamma) expressed.
Change in the cortical connectivity | Change from baseline to the end of treatment at week 24.
  Monitoring how TMS-induced EEG activity spreads from the stimulated area to the other areas, it is possible to assess the effective connectivity that area has with a widespread of network connected. So we calculate the source reconstruction, coherence between different areas and other connectivity indexes in the cortical oscillatory domain, i.e. Phase-locking Value (PLV) and Phase-amplitude coupling (PAC).
Change in Virtual Reality task performance. | Change from baseline to the end of treatment at week 24.
  The motor task will be assessed using the Gait Real-time Analysis Interactive Lab (GRAIL) system and a certified VR headset, measuring kinematic variables (walking speed in m/s and joint trajectories in degrees) and performance metrics (number of targets hit and reaction time in ms) under dual-task conditions.
Changes in the blood-based biomarkers | Change from baseline to the end of treatment at week 24.
  Plasma concentrations of Aβ42, Aβ40, P-tau217, glial fibrillary acidic protein (GFAP), neurofilament light chain (NfL), neurogranin, SNAP25 will be quantified using Single Molecule Array (Simoa) assays and reported in pg/mL.
Changes on MRI markers of regional gray matter atrophy and functional connectivity | Change from baseline to the end of treatment at week 24.
  Will measure changes in brain structure, tissue integrity, and atrophy, as well as changes in brain activity and blood flow using resting-state functional MRI (fRMI) and arterial spin labeling (ASL).

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Koch, Prof., Principal Investigator — IRCCS Santa Lucia Foundation
Locations (2):
- Italy (2):
  - IRCCS Santa Lucia Foundation, Rome, Italy
  - I.R.C.C.S. Centro Neurolesi Bonino Pulejo, Messina, Sicily

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou HY, Chen SC, Yen TH, Han HM. Effect of a Virtual Reality-Based Exercise Program on Fatigue in Hospitalized Taiwanese End-Stage Renal Disease Patients Undergoing Hemodialysis. Clin Nurs Res. 2020 Jul;29(6):368-374. doi: 10.1177/1054773818788511. Epub 2018 Jul 15. PMID 30009636
- [Background] Blennow K, Zetterberg H. Biomarkers for Alzheimer's disease: current status and prospects for the future. J Intern Med. 2018 Dec;284(6):643-663. doi: 10.1111/joim.12816. Epub 2018 Aug 19. PMID 30051512
- [Background] Fox MD, Halko MA, Eldaief MC, Pascual-Leone A. Measuring and manipulating brain connectivity with resting state functional connectivity magnetic resonance imaging (fcMRI) and transcranial magnetic stimulation (TMS). Neuroimage. 2012 Oct 1;62(4):2232-43. doi: 10.1016/j.neuroimage.2012.03.035. Epub 2012 Mar 19. PMID 22465297
- [Background] Gili T, Cercignani M, Serra L, Perri R, Giove F, Maraviglia B, Caltagirone C, Bozzali M. Regional brain atrophy and functional disconnection across Alzheimer's disease evolution. J Neurol Neurosurg Psychiatry. 2011 Jan;82(1):58-66. doi: 10.1136/jnnp.2009.199935. Epub 2010 Jul 16. PMID 20639384
- [Background] Koch G, Casula EP, Bonni S, Borghi I, Assogna M, Minei M, Pellicciari MC, Motta C, D'Acunto A, Porrazzini F, Maiella M, Ferrari C, Caltagirone C, Santarnecchi E, Bozzali M, Martorana A. Precuneus magnetic stimulation for Alzheimer's disease: a randomized, sham-controlled trial. Brain. 2022 Nov 21;145(11):3776-3786. doi: 10.1093/brain/awac285. PMID 36281767
- [Background] Koch G, Bonni S, Pellicciari MC, Casula EP, Mancini M, Esposito R, Ponzo V, Picazio S, Di Lorenzo F, Serra L, Motta C, Maiella M, Marra C, Cercignani M, Martorana A, Caltagirone C, Bozzali M. Transcranial magnetic stimulation of the precuneus enhances memory and neural activity in prodromal Alzheimer's disease. Neuroimage. 2018 Apr 1;169:302-311. doi: 10.1016/j.neuroimage.2017.12.048. Epub 2017 Dec 19. PMID 29277405
- [Background] Hu Y, Kirmess KM, Meyer MR, Rabinovici GD, Gatsonis C, Siegel BA, Whitmer RA, Apgar C, Hanna L, Kanekiyo M, Kaplow J, Koyama A, Verbel D, Holubasch MS, Knapik SS, Connor J, Contois JH, Jackson EN, Harpstrite SE, Bateman RJ, Holtzman DM, Verghese PB, Fogelman I, Braunstein JB, Yarasheski KE, West T. Assessment of a Plasma Amyloid Probability Score to Estimate Amyloid Positron Emission Tomography Findings Among Adults With Cognitive Impairment. JAMA Netw Open. 2022 Apr 1;5(4):e228392. doi: 10.1001/jamanetworkopen.2022.8392. PMID 35446396